CLINICAL TRIAL: NCT02561871
Title: Phase 1, First in Human Study to Evaluate the Safety, Tolerability and Immunogenicity of Ad26.RSV.FA2 Followed by Ad35.RSV.FA2 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of Ad26.RSV.FA2 Followed by Ad35.RSV.FA2 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR107705; VAC18192RSV1003 (Other: Crucell Holland BV)
Record Dates: First submitted 2015-08-21; First posted 2015-09-28 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Syncytial Viruses; Respiratory Tract Infections
Keywords: Ad26.RSV.FA2 (JNJ-61187165-AAA); Ad35.RSV.FA2 (JNJ-61187191-AAA); Healthy participants
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Two subsequent Intramuscular injections of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on Day 1 and Day 85, and one intramuscular injection of Ad35.RSV.FA2 (1x10^11 virus particles [vp]) on Day 169.
  Interventions: Biological: Ad26.RSV.FA2; Biological: Ad35.RSV.FA2
- Group 2 (Experimental): Intramuscular injection of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on Day 1, an intramuscular injection of Ad35.RSV.FA2 (1x10^11 vp) on Day 85 and and an intramuscular injection of placebo control consisting of the vaccine formulation buffer on Day 169.
  Interventions: Biological: Ad26.RSV.FA2; Biological: Ad35.RSV.FA2; Drug: Placebo
- Group 3 (Experimental): Three intramuscular injections of placebo control on Day 1, Day 85 and Day 169.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.FA2 — Participants will receive Intramuscular injection of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on day 1 and 85 in Group 1. Intramuscular injection of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on day 1 in Group 2.
  Other Names: JNJ-61187165-AAA
  Arms: Group 1; Group 2
Biological: Ad35.RSV.FA2 — Participants will receive Intramuscular injection of Ad35.RSV.FA2 (1x10^11 virus particles [vp]) on day 169 in Group 1. Intramuscular injection of Ad35.RSV.FA2 (1x10^11 virus particles [vp]) on day 85 in Group 2.
  Other Names: JNJ-61187191-AAA
  Arms: Group 1; Group 2
Drug: Placebo — Participants will receive Intramuscular injection of Placebo control on day 169 in Group 2. Intramuscular injection of Placebo control on day 1, 85 and 169 in Group 3.
  Arms: Group 2; Group 3

SUMMARY:
The purpose of this study is to assess the safety and tolerability of intramuscular prime-boost regimens of Ad26.RSV.FA2 given either once or twice followed by Ad35.RSV.FA2 (human adenovirus-vectored vaccine candidate) in healthy participants.

DETAILED DESCRIPTION:
This is a single-center, randomized (study vaccine assigned to participants by chance), placebo-controlled study (an inactive substance; a pretend treatment [with no vaccine in it] that is compared in a clinical trial with a vaccine to test if the vaccine has a real effect), double-blind (neither the researchers nor the participants know what treatment the participant is receiving) Phase 1 study in healthy participants. The study comprises a 4-week screening period; vaccination for each participant on Days 1, 85, and, 169; a 28-day follow-up period performed after each vaccination and a final visit at Day 337. Approximately 32 Participants will be randomized in parallel in a 3:3:2 ratio to 3 treatment groups (Group 1/2/3) to receive either Ad26.RSV.FA2 or Ad35.RSV.FA2 or placebo. The study duration will be approximately 52 weeks. Blood samples for immunogenicity will be collected. Participant's safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be in good health, without significant medical illness, on the basis of physical examination, medical history, vital signs measurement, and 12-lead electrocardiogram (ECG) performed at screening
* Participant must meet protocol defined laboratory criteria within 28 days before Day 1
* Before randomization, a woman must be either; Not of childbearing potential: postmenopausal or surgically sterilized; of childbearing potential and practicing an effective method of birth control before vaccination and through 3 months after the last vaccination. Women, who are not heterosexually active at screening, must agree to utilize highly-effective method of birth control if they become heterosexually active until 3 months after receiving the last dose of study vaccine
* A woman must have a negative serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at the screening visit, and a negative urine pregnancy test pre-vaccination on Day 1
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction until 3 months after receiving the last dose of study vaccine. A man must agree not to donate sperm until 3 months after receiving the last dose of study vaccine

Exclusion Criteria:

* Participant has a body mass index (BMI) less than or equal to (<=)19 and greater than or equal to (>=30) kilogram per square meter (kg/m2)
* Participant has any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude participation (e.g. history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, poorly controlled asthma, active tuberculosis or other systemic infections)
* Participant has had major surgery within the 4 weeks prior to randomization or has planned major surgery through the course of the study
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Participant has human immunodeficiency virus (HIV) type 1 or type 2 infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) | Up to 8 days after each vaccination
  Solicited AEs are precisely defined events that participants are specifically asked about and which are noted by participants through the participant diary.
Number of Participants with Solicited Systemic Adverse Events (AEs) | Up to 8 days after each vaccination
Number of Participants with Unsolicited AEs | From Signing of informed consent up to 28 days after each vaccination
  Unsolicited AEs will be reported by the participant from when the informed consent form (ICF) is signed until 28 days after each vaccination, or early discontinuation.
Number of Participants with Serious Adverse Events (SAEs) | From Signing of informed consent up to Day 337
  A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens as Measured by a Virus Neutralization Assay | Day 1 (predose) up to day 337
Immune Responses to the Study Vaccine Regimens Measured by an Enzyme-linked Immunosorbent Assay (ELISA) | Day 1 (predose) up to day 337
Immune responses to the study vaccine regimens as measured by an Enzyme-linked Immunospot Assay (ELISpot) | Day 1 (predose) up to day 337
  Enzyme-linked Immunospot Assay (ELISpot) is used to quantify the amount of peripheral blood mononuclear cells (PBMCs) able to produce Interferon-gamma upon RSV antigen stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (1):
- Miami, Florida, United States